CLINICAL TRIAL: NCT00931554
Title: Early Versus Standard Drainage Removal After Pancreatic Resections: Results of a Prospective Randomized Clinical Trial
Brief Title: Randomized Trial of Early Versus Standard Drainage Removal After Pancreatic Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Claudio Bassi MD, Professor of Surgery, Department of Surgical and Gastroenterological Sciences, University of Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DREN-01
Record Dates: First submitted 2009-05-28; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Pancreaticoduodenectomy; Distal Pancreatectomy; Pancreatic Fistula; Abdominal Abscess
MeSH Terms: conditions — Pancreatic Fistula; Abdominal Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early drain removal (Active Comparator): Drain removal in postoperative day 3
  Interventions: Procedure: Postoperative drain removal
- Standard drain removal (Active Comparator): Drain removal on postoperative day 5
  Interventions: Procedure: Postoperative drain removal

INTERVENTIONS:
Procedure: Postoperative drain removal — removal of postoperative drainages at different time points (postoperative day 3 versus postoperative day 5)

SUMMARY:
Despite a substantial decrease in postoperative mortality, morbidity after pancreatic resections is still high, even at high-volume centers. It has been recently suggested that early removal of postoperative drainages is associated to a decreased rate of intra-abdominal complications, with particular regard to pancreatic fistula. Furthermore, our research group demonstrated that measuring amylase value in drainages (AVD) on postoperative day 1 plays a cardinal role in predicting the developement of abdominal complications, including pancreatic fistula. In particular, patients with an AVD lower than 5000 IU/L in postoperative day 1 were considered at low risk of fistula. Therefore, the investigators designed a randomized prospective trial on early (postoperative day 3) versus standard (postoperative day 5) drainages removal after pancreatic resections in patients at low risk of developing pancreatic fistula (AVD < 5000 IU/L in postoperative day 1) to test whether drainages "per se" influence postoperative complication rates and to eventually validate a fast-track policy in pancreatic resections.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone either pancreaticoduodenectomy (reconstruction by pancreaticojejunostomy) or distal pancreatectomy with an amylase value in drains on postoperative day 1 less than 5000 IU/L

Exclusion Criteria:

* Pancreaticoduodenectomy reconstructed with pancreaticogastrostomy
* Clinical suspect of postoperative haemorrhage within 72hours after the operation
* Clinical suspect of biliary fistula
* Fluid collection greater than 3cm at an ultrasound carried out on postoperative day 3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-03; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Abdominal Complications | 1 month

SECONDARY OUTCOMES:
In-hospital stay | 1 month
Pulmonary complications | 1 month
Hospital readmission | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery B, Policlinico G.B. Rossi, Verona, Italy

REFERENCES:
- [Background] Molinari E, Bassi C, Salvia R, Butturini G, Crippa S, Talamini G, Falconi M, Pederzoli P. Amylase value in drains after pancreatic resection as predictive factor of postoperative pancreatic fistula: results of a prospective study in 137 patients. Ann Surg. 2007 Aug;246(2):281-7. doi: 10.1097/SLA.0b013e3180caa42f. PMID 17667507
- [Background] Kawai M, Tani M, Terasawa H, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Yamaue H. Early removal of prophylactic drains reduces the risk of intra-abdominal infections in patients with pancreatic head resection: prospective study for 104 consecutive patients. Ann Surg. 2006 Jul;244(1):1-7. doi: 10.1097/01.sla.0000218077.14035.a6. PMID 16794381
- [Derived] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661